CLINICAL TRIAL: NCT03805191
Title: A Multicentre Observational Study to Investigate the Improvement in Glucose FLuctuation of Sufficient Acarbose Therapy on Type 2 Diabetes Patient With High Blood Glucose Fluctuation
Brief Title: A Study for Sufficient Acarbose Decreased Glucose Excursion in Type 2 Diabetic Patients
Acronym: FLAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: RD-OI-1257
Record Dates: First submitted 2019-01-10; First posted 2019-01-15 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes Mellitus; Poor Glycemic Control
Keywords: Glycemic excursions; Acarbose; Continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicentre observational study to investigate the improvement in glucose fluctuation of sufficient acarbose therapy on type 2 diabetes patient with high blood glucose fluctuation

DETAILED DESCRIPTION:
Acarbose competitively inhibits the a-glycosidase on the surface of epithelial cells from the duodenum and small intestine, delays the metabolism and assimilation of carbohydrates, and thus effectively decreases postprandial blood glucose(PBG) as well as the risk of hypoglycemia before the next meal.Acarbose is now used as the preferred drug for some patients with prediabetes and newly diagnosed type 2 diabetes millitus(T2DM).This study aims to investigate the glycemic excursions with different courses and glycated hemoglobin A1c(HbA1c) levels after treated three months with acarbose.To minimize gastrointestinal side effects，starting dosage of acarbose of 50 mg is given orally three times daily for 10 days(with the first bite) of each main meal. Glycemic excursions are evaluated using the mean amplitude of glycemic excursions (MAGE), the postprandial glycemic excursions (PPGE) and the largest amplitude of glycemic excursions (LAGE).Freestyle Libre flash glucose monitoring system (FGMS，Abbott Laboratories,USA) was administered in this study. According to the standard Freestyle Libre Pro operating guidelines, the FGMS is installed in all participants to monitor glucose levels of interstitial fluid for 14 consecutive days. The glucose sensor is inserted into the subcutaneous tissue of upper arm at 8:00-9:00 in the morning.Glucose concentrations at 7 preset times per day (before meals, 2-h after meals and at bedtime) were determined with VivaChek Ino Smart（VivaChek Laboratories, Inc., USA) every two weeks.Four days before using acarbose and five weeks after using acarbose, FGMS was using to monitor the continuous glucose.MAGE was calculated for each subject by taking the arithmetic mean of FGM values increased or decreased (from nadirs to peaks or vice versa) when both ascending and descending segments exceeded the value of one standard deviation (SD) of the FGM values for 24-h period.The primary endpoint of the study is the extent of change in MAGE.Secondary endpoints are changes in PPGE,LAGE and HbA1c. Gene polymorphism is detected for enrolled patient with poor acarbose effect.

ELIGIBILITY:
Inclusion Criteria:

1. All enrolled patients sign the informed consent. sign the informed consent form.
2. Clinical diagnosis of T2DM(1999 WHO).
3. No acarbose in nearly 3 months.
4. 7% < HbA1c ≤10% .
5. PPGE >2.2mmol/L and LAGE >4.4mmol/L.
6. MAGE > 3.9 mmol/L.
7. The previous therapy remain the same.
8. Contraception is needed for women of child-bearing age until 28 days after the end.

Exclusion Criteria:

1. Women of childbearing potential unable or unwilling to use acceptable birth control, or women who are pregnant or breastfeeding.
2. Replacement or chronic systemic corticosteroid therapy. Cytochrome P450 3A4 enzyme inducer or inhibitor therapy.Antiviral therapy for immunodeficiency disease.
3. History of gastrointestinal disease or surgery including Roemheld Syndrome, severe hernia, intestinal obstruction, intestinal ulcer, gastroenterostomy, enterectomy, bariatric surgery or lap-band procedure.
4. Known immunocompromised status, including but not limited to, individuals who had undergone organ transplantation or acquired immunodeficiency syndrome (AIDS).
5. History of hemoglobinopathy .
6. Any subject who was currently abusing alcohol or other drugs or had done so within the last 12 months.
7. There are contraindications listed in the acarbose instructions.
8. History of acute or chronic pancreatitis, or current acute or chronic pancreatitis.
9. Type 1 diabetees mellitus.
10. History of diabetic ketoacidosis or hyperosmolar nonketosis coma in recent 1 month.
11. Patients with clinically apparent hepatobiliary disease, including but not limited to chronic active hepatitis and/or severe hepatic insufficiency. Alanine Aminotransferase(ALT) or Aspartate Aminotransferase(AST) > 3x upper limit of normal (ULN), or serum total bilirubin (TB) >34.2 μmol/L (>2 mg/dL).
12. Patients with following renal disease history or renal disease related features:

    1. History of unstable or rapidly progressing renal disease;
    2. Patients with moderate /severe renal impairment or end-stage renal disease (eGFR< 60 mL/min/1.73 m2);
    3. Urinary albumin: creatinine ratio >1800 mg/g;
    4. Serum creatinine (Cr) ≥133 μmol/L (≥1.50 mg/dL) for male subjects; Serum Cr≥124 μmol/L (≥1.40 mg/dL) for female subjects;
    5. Conditions of congenital renal glycosuria.
13. Any of the following cardiovascular diseases within 6 months of the enrollment visit:

    1. Myocardial infarction;
    2. Cardiac surgery or revascularization (coronary artery bypass graft/percutaneous transluminal coronary angioplasty);
    3. Unstable angina;
    4. Congestive heart failure New York Heart Association Class III or IV;
    5. Transient ischemic attack or significant cerebrovascular disease.
14. Any subject , in the judgment of the investigator, was at risk that might affect the interpretation of efficacy or safety data or the conduct ion of the study，including laboratory and physical examination or ECG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the course of diabetes, enrolled patients are divided into three groups: A (< 5Y), B (5-10y), C (> 10Y). According to the level of HbA1c,enrolled patients are divided into three groups:I (7%-8%), II (8%-9%), and III (9%-10%). Then there are nine groups, namely AI, AII, AIII, BI, BII, BIII, CI, CII, and CIII.100 patients are enrolled in each group.All enrolled patiens are 900.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The extent of change in MAGE | 8 weeks
  Mean absolute glucose excursions (MAGE) was calculated to assess intraday glucose variability. The difference between the consecutive peaks and nadirs exceeding one standard deviation (SD) of the daily mean blood glucose (MBG) level was expressed as absolute glucose excursion (AGE). MAGE was an arithmetic mean of all absolute AGEs.The average MAGE of the last three days of the eighth week are compared with the baseline（The average MAGE of the three days before using acarbose).The extent of change in MAGE is numerical value to to assess glucose variability.

SECONDARY OUTCOMES:
The extent of change in PPGE,LAGE | 8 weeks
  Postprandial glucose excursion (PPGE) is calculated as the peak value of glucose after meals minus the glucose level at the beginning of each meal to evaluate the influence of meals on glucose fluctuation.Largest amplitude of glycemic excursions (LAGE) is calculated as the maximum minus the minimum blood glucose levels measured in one day.The average PPGE、LAGE of the last three days of the eighth week compared with the baseline（The average PPGE、LAGE of the three days before using acarbose）.
The control rate of HbA1c | 12 weeks
  When HbA1c<7% was considered as the criteria, the control rate of HbA1c after 12 weeks.

OTHER OUTCOMES:
Gene polymorphism | 12 weeks
  Gene polymorphism is detected for enrolled patient with poor acarbose effect.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Liao, MD, Principal Investigator — Qianfoshan Hospital; Yuping Zhou, MD, Principal Investigator — Weihai Municipal Hospital; Shuguang Pang, MD, Principal Investigator — Jinan Central Hospital; Fei Wang, MD, Principal Investigator — Huangdao Branch of Affiliated Hospital of Medical College,Qingdao University; Yongjun Jin, MD, Principal Investigator — Yantai Branch of Affiliated Binzhou Medical College; Tianying Xu, MD, Principal Investigator — People's hospital of Qihe county; Guangzhen Zhang, MD, Principal Investigator — Liaocheng People's Hospital; Yunfeng Zhang, MD, Principal Investigator — Linyi lanshan district diabetes hospital; Lin Sun, MD, Principal Investigator — Jining Medical University; Dadong Fei, MD, Principal Investigator — Zaozhuang Municipal Hospital; Guangling Xu, MD, Principal Investigator — Guanxian people's hospital of liaocheng city
Locations (1):
- Qilu Hospital of Shandong University, Jinan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xu Y, Wang L, He J, Bi Y, Li M, Wang T, Wang L, Jiang Y, Dai M, Lu J, Xu M, Li Y, Hu N, Li J, Mi S, Chen CS, Li G, Mu Y, Zhao J, Kong L, Chen J, Lai S, Wang W, Zhao W, Ning G; 2010 China Noncommunicable Disease Surveillance Group. Prevalence and control of diabetes in Chinese adults. JAMA. 2013 Sep 4;310(9):948-59. doi: 10.1001/jama.2013.168118. PMID 24002281
- [Background] Poolsup N, Suksomboon N, Rattanasookchit S. Meta-analysis of the benefits of self-monitoring of blood glucose on glycemic control in type 2 diabetes patients: an update. Diabetes Technol Ther. 2009 Dec;11(12):775-84. doi: 10.1089/dia.2009.0091. PMID 20001678
- [Background] The relationship of glycemic exposure (HbA1c) to the risk of development and progression of retinopathy in the diabetes control and complications trial. Diabetes. 1995 Aug;44(8):968-83. PMID 7622004
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Monnier L, Colette C, Dunseath GJ, Owens DR. The loss of postprandial glycemic control precedes stepwise deterioration of fasting with worsening diabetes. Diabetes Care. 2007 Feb;30(2):263-9. doi: 10.2337/dc06-1612. PMID 17259492
- [Background] Maia FF, Araujo LR. Efficacy of continuous glucose monitoring system (CGMS) to detect postprandial hyperglycemia and unrecognized hypoglycemia in type 1 diabetic patients. Diabetes Res Clin Pract. 2007 Jan;75(1):30-4. doi: 10.1016/j.diabres.2006.05.009. Epub 2006 Jun 27. PMID 16806560
- [Background] Mastrototaro J. The MiniMed Continuous Glucose Monitoring System (CGMS). J Pediatr Endocrinol Metab. 1999;12 Suppl 3:751-8. No abstract available. PMID 10626266
- [Background] Ginsberg BH. The FDA panel advises approval of the first continuous glucose sensor. Diabetes Technol Ther. 1999 Summer;1(2):203-4. doi: 10.1089/152091599317431. No abstract available. PMID 11475294
- [Background] Monnier L, Colette C, Owens DR. Glycemic variability: the third component of the dysglycemia in diabetes. Is it important? How to measure it? J Diabetes Sci Technol. 2008 Nov;2(6):1094-100. doi: 10.1177/193229680800200618. PMID 19885298
- [Background] Guerci B. [Asymptomatic glycemic instability: how to measure it and which clinical applications? ]. Diabetes Metab. 2003 Apr;29(2 Pt 1):179-88. French. PMID 12746641
- [Background] Hirsch IB, Brownlee M. Should minimal blood glucose variability become the gold standard of glycemic control? J Diabetes Complications. 2005 May-Jun;19(3):178-81. doi: 10.1016/j.jdiacomp.2004.10.001. PMID 15866065
- [Background] Del Prato S. In search of normoglycaemia in diabetes: controlling postprandial glucose. Int J Obes Relat Metab Disord. 2002 Sep;26 Suppl 3:S9-17. doi: 10.1038/sj.ijo.0802172. PMID 12174318
- [Background] Yang W, Liu J, Shan Z, Tian H, Zhou Z, Ji Q, Weng J, Jia W, Lu J, Liu J, Xu Y, Yang Z, Chen W. Acarbose compared with metformin as initial therapy in patients with newly diagnosed type 2 diabetes: an open-label, non-inferiority randomised trial. Lancet Diabetes Endocrinol. 2014 Jan;2(1):46-55. doi: 10.1016/S2213-8587(13)70021-4. Epub 2013 Oct 18. PMID 24622668
- [Background] Li S, Xiao J, Ji L, Weng J, Jia W, Lu J, Zhou Z, Guo X, Liu J, Shan Z, Zhu D, Chen L, Zhao Z, Tian H, Ji Q, Ge J, Li Q, Lin L, Yang Z, He J, Yang W; China National Diabetes and Metabolic Disorders Study Investigators. BMI and waist circumference are associated with impaired glucose metabolism and type 2 diabetes in normal weight Chinese adults. J Diabetes Complications. 2014 Jul-Aug;28(4):470-6. doi: 10.1016/j.jdiacomp.2014.03.015. Epub 2014 Apr 1. PMID 24809931
- [Background] Ma RC. Acarbose: an alternative to metformin for first-line treatment in type 2 diabetes? Lancet Diabetes Endocrinol. 2014 Jan;2(1):6-7. doi: 10.1016/S2213-8587(13)70107-4. Epub 2013 Oct 18. No abstract available. PMID 24622656
- [Background] Chen M, Dou J, Zhuang X, Dong L, Ruan D, Ding J, Zhang Y, Tian Y, Zhao J, Wu J, Fu Y, Huang X, Wang S, Lu J. [An analysis of hypoglycemic agents used among patients with type 2 diabetes in Beijing communities]. Zhonghua Nei Ke Za Zhi. 2014 Feb;53(2):112-5. Chinese. PMID 24767162
- [Background] Ju-Ming L, Xiao-Hui G, Xiao-Feng L, Yan-Bing L, Li Y, Yao-Ming X. Effects of Nateglinide on Postprandial Plasma Glucose Excursion and Metabolism of Lipids in Chinese Patients with Type 2 Diabetes：A 4-week, randomized, active-control, open-label, parallel-group, multicenter trial. Curr Med Res Opin. 2012 Jul 19. doi: 10.1185/03007995.2012.713340. Online ahead of print. PMID 22809112
- [Background] Zhou J, Li H, Zhang X, Peng Y, Mo Y, Bao Y, Jia W. Nateglinide and acarbose are comparably effective reducers of postprandial glycemic excursions in chinese antihyperglycemic agent-naive subjects with type 2 diabetes. Diabetes Technol Ther. 2013 Jun;15(6):481-8. doi: 10.1089/dia.2013.0046. Epub 2013 Apr 30. PMID 23631607
- [Background] Wang JS, Lin SD, Lee WJ, Su SL, Lee IT, Tu ST, Tseng YH, Lin SY, Sheu WH. Effects of acarbose versus glibenclamide on glycemic excursion and oxidative stress in type 2 diabetic patients inadequately controlled by metformin: a 24-week, randomized, open-label, parallel-group comparison. Clin Ther. 2011 Dec;33(12):1932-42. doi: 10.1016/j.clinthera.2011.10.014. Epub 2011 Nov 10. PMID 22078152
- [Background] Lin SD, Wang JS, Hsu SR, Sheu WH, Tu ST, Lee IT, Su SL, Lin SY, Wang SY, Hsieh MC. The beneficial effect of alpha-glucosidase inhibitor on glucose variability compared with sulfonylurea in Taiwanese type 2 diabetic patients inadequately controlled with metformin: preliminary data. J Diabetes Complications. 2011 Sep-Oct;25(5):332-8. doi: 10.1016/j.jdiacomp.2011.06.004. Epub 2011 Aug 2. PMID 21813293
- [Background] Nomoto H, Miyoshi H, Sugawara H, Ono K, Yanagiya S, Oita M, Nakamura A, Atsumi T. A randomized controlled trial comparing the effects of dapagliflozin and DPP-4 inhibitors on glucose variability and metabolic parameters in patients with type 2 diabetes mellitus on insulin. Diabetol Metab Syndr. 2017 Jul 17;9:54. doi: 10.1186/s13098-017-0255-8. eCollection 2017. PMID 28725273
- [Background] Makdissi A, Chaudhuri A, Kuhadiya N, Batra M, Dandona P. Comment on: Rizzo et al. Reduction of oxidative stress and inflammation by blunting daily acute glucose fluctuations in patients with type 2 diabetes: role of dipeptidyl peptidase-IV inhibition. Diabetes Care 2012;35:2076-2082. Diabetes Care. 2013 Jun;36(6):e80. doi: 10.2337/dc12-2220. No abstract available. PMID 23704688
- [Background] Polidori D, Sha S, Mudaliar S, Ciaraldi TP, Ghosh A, Vaccaro N, Farrell K, Rothenberg P, Henry RR. Canagliflozin lowers postprandial glucose and insulin by delaying intestinal glucose absorption in addition to increasing urinary glucose excretion: results of a randomized, placebo-controlled study. Diabetes Care. 2013 Aug;36(8):2154-61. doi: 10.2337/dc12-2391. Epub 2013 Feb 14. PMID 23412078
- [Background] Deshmukh AB, Patel MC, Mishra B. SGLT2 inhibition: a novel prospective strategy in treatment of diabetes mellitus. Ren Fail. 2013;35(4):566-72. doi: 10.3109/0886022X.2013.766560. Epub 2013 Feb 25. PMID 23438184
- [Background] Wu H, Liu J, Lou Q, Liu J, Shen L, Zhang M, Lv X, Gu M, Guo X. Comparative assessment of the efficacy and safety of acarbose and metformin combined with premixed insulin in patients with type 2 diabetes mellitus. Medicine (Baltimore). 2017 Sep;96(35):e7533. doi: 10.1097/MD.0000000000007533. PMID 28858080
- [Background] Wang JS, Lee IT, Lee WJ, Lin SD, Su SL, Tu ST, Tseng YH, Lin SY, Sheu WH. Glycemic excursions are positively associated with HbA1c reduction from baseline after treatment with acarbose in patients with type 2 diabetes on metformin monotherapy. J Diabetes. 2017 Mar;9(3):248-255. doi: 10.1111/1753-0407.12406. Epub 2016 May 31. PMID 27043224
- [Background] Park S, Choi SB. Induction of long-term normoglycemia without medication in Korean type 2 diabetes patients after continuous subcutaneous insulin infusion therapy. Diabetes Metab Res Rev. 2003 Mar-Apr;19(2):124-30. doi: 10.1002/dmrr.343. PMID 12673780
- [Background] Naqvi S, Naveed S, Ali Z, Ahmad SM, Asadullah Khan R, Raj H, Shariff S, Rupareliya C, Zahra F, Khan S. Correlation between Glycated Hemoglobin and Triglyceride Level in Type 2 Diabetes Mellitus. Cureus. 2017 Jun 13;9(6):e1347. doi: 10.7759/cureus.1347. PMID 28713663